CLINICAL TRIAL: NCT01246245
Title: Nursing Care Management of External Fixation in Hospitalization: Pin Site Infection Incidence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr AMI MAYO, Rambam Health Care Campus
Other Study IDs: 049-10 CTIL
Record Dates: First submitted 2010-11-21; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-07

CONDITIONS: Infection
Keywords: PIN SITE INFECTION AFTER EXTERNAL FIXATION
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The incidence of pin site infection is related to the nursing management of external fixation.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old patients

Exclusion Criteria:

* Immune Depression
* Patients who are treated with immunosupressive drugs or steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after external fixation insertion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-12

PRIMARY OUTCOMES:
Pin Site Infection Incidence | 6 MONTH